CLINICAL TRIAL: NCT02728921
Title: The Importance of Albumin Infusion Rate for Plasma Volume Expansion. AIR. A Phase III Assessor Blinded Parallel Group Randomized Study
Brief Title: The Importance of Albumin Infusion Rate for Plasma Volume Expansion Following Major Abdominal Surgery
Acronym: AIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-004446-42
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Neoplasms; Urogenital Neoplasm; Systemic Inflammatory Response Syndrome; Hypovolemia
MeSH Terms: conditions — Pancreatic Neoplasms; Urogenital Neoplasms; Systemic Inflammatory Response Syndrome; Hypovolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% Albumin infusion 30 min (Active Comparator): Intravenous infusion of 5% Albumin at a dose of 10ml/kg during 30 min.
  Interventions: Drug: 5% Albumin infusion 30 min
- 5% Albumin infusion 3 hours (Experimental): Intravenous infusion of 5% Albumin at a dose of 10ml/kg during 3 hours. Dose is based on ideal body weight
  Interventions: Drug: 5% Albumin infusion 3 hours

INTERVENTIONS:
Drug: 5% Albumin infusion 30 min — Intravenous infusion of 5% Albumin at a dose of 10 ml/kg during 30 minutes. Dose is based on ideal weight.
  Arms: 5% Albumin infusion 30 min
Drug: 5% Albumin infusion 3 hours — Intravenous infusion of 5% Albumin at a dose of 10 ml/kg during 3 hours. Dose is based on ideal weight.
  Arms: 5% Albumin infusion 3 hours

SUMMARY:
To study if plasma volume expansion is influenced by the rate at which a colloidal solution is administered in patients with a systemic inflammatory response induced by major abdominal surgery.

Randomization will be performed postoperatively at the day of surgery with a 1:1 ratio with no stratification and the study drug will be given as a slow (3 hours) or rapid (30 minutes) intravenous infusion.

DETAILED DESCRIPTION:
Major surgery is one of many triggers of a systemic inflammatory response syndrome (SIRS), which disrupts the normal regulation of transcapillary fluid exchange with tissue oedema and hypovolemia as a consequence. Hypovolemia will amplify the inflammatory reaction by reducing cardiac output and oxygen delivery, which creates a vicious circle. Fluid therapy is therefore a cornerstone in the perioperative treatment patients subjected to major surgery. However, even if fluid therapy is life saving it is also associated with side effects such as further oedema formation, coagulopathy and further endothelial dysfunction.

From a clinical perspective, it is therefore important that the fluid administered to antagonize hypovolemia as far as possible remains intravascularly. Colloids are macromolecules for which the vessel wall has a low permeability and proponents of colloid containing fluids argues that less volume is required for equal plasma volume compared to crystalloids. However, extravasation of colloids is not only a function of the vessel wall permeability but is also dependent on the volume of fluid to that is filtered across the vascular wall, which in turn depends on the trans-capillary hydrostatic pressure. This means that administration of colloids in a way that minimizes the increase in capillary pressure could be important for the plasma volume expanding effect.

In support of this hypothesis is the experimental result that the plasma volume expansion of a colloidal solution can be affected by the rate of administration (Bark et al., 2013). If this finding proves to be valid also in a clinical setting, it will be very important for how colloidal solutions are prescribed in the clinic and may change current clinical practice in which suspected hypovolemia often is treated with a bolus infusion of fluid. This study intend to investigate whether these findings can be reproduced after a so-called Whipple's operation or after major gynaecological cancer surgery.

Study patients will be studied after these procedures because because they are large and standardized operations that trigger an inflammatory condition with capillary leakage and therefore can be considered as a model for major surgical procedures as well as ICU patients with SIRS triggered by for example sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is scheduled for non-emergent Whipple operation or major gynaecological cancer surgery.
2. Indication for fluid therapy as judged by the anaesthesiologist in charge and at least one at least one of the following criteria is fulfilled:

   * Positive "leg raising test" (pulse pressure increase > 9% or stroke volume increase by more than 10% as measured with cardiac ultrasound.
   * Central venous oxygen saturation (ScvO2) < 70%.
   * Plasma lactate > 2.0 mmol/l.
   * Urine output < 0.5 ml / kg for the latest hour.
   * Respiratory variation of the inferior vena cava of more than 15% as measured by ultrasound.
   * Systolic pressure < 100 mmHg, mean arterial pressure < 55 mmHg
3. Age 40 and above
4. Written consent by patient to participate in the study

Exclusion Criteria:

1. Hypersensitivity to the active drug/ the tracer.
2. Signs of postoperative bleeding.
3. History of heart failure.
4. The responsible physician considers that there are strong reasons to administrate another fluid or same fluid but in another way or in a different volume than those included in the protocol.
5. Pregnancy
6. Clinical judgment by the investigator or the treating physician that the patient should not participate in of the study for reasons other than described above.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in plasma volume | From start of infusion until 3 hours after start of infusion

SECONDARY OUTCOMES:
Change in plasma volume over time | From start of infusion until 3 hours after start of infusion
  Integral of plasma volume over time
Incidence of postoperative complications | 30 days postoperatively

OTHER OUTCOMES:
Transcapillary escape rate (TER) for albumin | 180-240 min after start of infusion
Change in heart rate, change in central venous oxygen saturation, change in haemoglobin concentration in blood, change in blood pressure, change in central venous pressure, change in plasma lactate and diuresis. | From start of infusion until 3 hours after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data collected in the current study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Statkevicius S, Bonnevier J, Bark BP, Larsson E, Oberg CM, Kannisto P, Tingstedt B, Bentzer P. The importance of albumin infusion rate for plasma volume expansion following major abdominal surgery - AIR: study protocol for a randomised controlled trial. Trials. 2016 Dec 7;17(1):578. doi: 10.1186/s13063-016-1714-5. PMID 27923389